CLINICAL TRIAL: NCT01669213
Title: Effects of Different Kinds, Different Doses of 5-HT3 Receptor Antagonists on Prevention of Hypotension After Spinal Anesthesia
Brief Title: Effects of Different Kinds, Different Doses of 5-HT3 Receptor Antagonists on Prevention of Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonsik Ahn, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: WSAhn_ramosetron_hypotension
Record Dates: First submitted 2012-08-10; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Hypotension; Shivering; Nausea and Vomiting; Vasopressor
Keywords: 5-HT3 receptor antagonist; hypotension; spinal anesthesia
MeSH Terms: conditions — Hypotension; Nausea; Vomiting | interventions — ramosetron; Ondansetron

ARMS (4):
- ramosetron 0.3 mg (Active Comparator): preparation of ramosetron 0.3 mg
  Interventions: Drug: ramosetron
- ondansetron 8 mg (Active Comparator): preparation of ondansetron 8mg
  Interventions: Drug: ondansetron
- ondansetron 4 mg (Active Comparator): preparation of ondansetron 4mg
  Interventions: Drug: ondansetron
- non 5-HT3 receptor antagonist (Placebo Comparator): preparation of normal saline 5 ml
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ramosetron — before 5 minutes spinal anesthesia, injection of ramosetron 0.3 mg
  Arms: ramosetron 0.3 mg
Drug: ondansetron — before 5 minutes spinal anesthesia, injection of ondansetron 8 mg
  Arms: ondansetron 8 mg
Drug: ondansetron — before 5 minutes spinal anesthesia, injection of ondansetron 4 mg
  Arms: ondansetron 4 mg
Drug: placebo — before 5 minutes spinal anesthesia, injection of normal saline 5 ml
  Arms: non 5-HT3 receptor antagonist

SUMMARY:
The purpose of this study is to estimate effects of different kinds, different dose of 5-HT3 receptor antagonists on prevention of hypotension after spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing spinal anesthesia

Exclusion Criteria:

* hypersensitivity on 5-HT3 receptor antagonists hypertension cardiovascular disease intake of selective serotonin reuptake inhibitor

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
prevention of hypotension by calcaulation the gap between baseline mean arterial pressure and lowest mean arterial pressure measured during 30 minutes after spinal anesthesia. | up to 30mins after spinal anesthesia
  comparasion of significantly difference in the gap between baseline mean arterial pressure and lowest mean arterial pressure measured during 30 minutes after spinal anesthesia.

SECONDARY OUTCOMES:
prevention of hypotension bycalculation the gap baseline systolic and diastolic blood pressure and lowerst systolic and diastolic blood pressure | up to 30mins after spinal anesthesia
  comparasion of significantly difference in the gap between baseline systolic arterial pressure and lowest systolic arterial pressure measured during 30 minutes after spinal anesthesia and the gap between baseline diastolic arterial pressure and lowest diastolic arterial pressure measured during 30 minutes after spinal anesthesia.

OTHER OUTCOMES:
occurrence ratio of shivering, nausea and vomiting, and usage doses of vasopressor (ephedrine or phenylephrine), and atropine | up to 30 min after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea